CLINICAL TRIAL: NCT03346681
Title: N-Acetyl-cysteine in Early Acute Respiratory Distress Syndrome
Acronym: NARDS
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no patients enrolled
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PalmettoHealth
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Patients meeting inclusion criteria will be randomly assigned to the treatment or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NAC and albuterol (Experimental): The procedure involved would be the administration of N-acetylcysteine via nebulization, which would be administered to the patient by respiratory therapy in the dosage of 2 mL 20% solution acetylcysteine (or 4 mL of 10% solution) along with inhaled albuterol via endotracheal tube every six hours for 72 hours total. The control arm will have saline administered with the albuterol every six hours. Both arms will have additional bronchodilators administered as indicated clinically (bronchospasm, COPD, peak airway pressure elevation, etc.).
  Interventions: Drug: N-acetyl cysteine
- Albuterol (No Intervention): Albuterol will be administered via nebulization every six hours.

INTERVENTIONS:
Drug: N-acetyl cysteine — The procedure involved would be the administration of N-acetylcysteine via nebulization, which would be administered to the patient by respiratory therapy in the dosage of 2 mL 20% solution acetylcysteine (or 4 mL of 10% solution) along with inhaled albuterol via endotracheal tube every six hours for 72 hours total. The control arm will have saline administered with the albuterol every six hours. Both arms will have additional bronchodilators administered as indicated clinically (bronchospasm, COPD, peak airway pressure elevation, etc.).
  Arms: NAC and albuterol

SUMMARY:
We would study whether there is any measurable benefit of the administration of nebulized n-acetyl-cysteine to acute respiratory distress syndrome patients starting within 48 hours of intubation and mechanical ventilation.

DETAILED DESCRIPTION:
Objectives / Research Aims The overall objectives of this study are to demonstrate whether a protocol for the early use of inhaled N-acetylcysteine improves mortality, ventilator days, ICU days, hospital stay, as well as the need for other "rescue" modalities, such as use of advanced ventilator modalities (such as airway pressure release ventilation [APRV]), paralytics, and prone positioning. As this is a pilot study, we would address the feasibility of recruiting and consenting patients as well as to ascertain the sample size that would be needed to power the desired endpoints in a larger study.

Setting The project will be performed in the Medical Intensive Care Unit at Palmetto Health Richland using subjects with severe acute respiratory distress syndrome that are identified within 48 hours of their disease process.

Resources Available It is not uncommon for the patients admitted with or that develop acute respiratory distress syndrome to receive breathing treatments of some variety, such as bronchodilators. This study would take an existing practice and add a relatively inexpensive medication, N-acetylcysteine.

It will be straightforward and require relatively little time to calculate the metrics for the patients enrolled in this study as these data are typically collected for intensive care unit patients already.

Our respiratory therapists are already very experienced and proficient at the administration of inhaled N-acetylcysteine. Likewise, the academic intensive care team would be able to readily classify the patients that are appropriate for this study as the partial pressure of oxygen to fraction of inspired oxygen (P/F) ratio is typically documented for every ventilated patient admitted to our unit.

Study Design Recruitment Methods The patients will be recruited based upon their P/F ratio less than 150 and being mechanically ventilated with a positive end expiratory pressure of 5 or greater. These patients will be started on the protocol within 48 hours of developing acute respiratory distress syndrome.

Inclusion and Exclusion Criteria Inclusion criteria includes adult patients admitted to the medical intensive care unit or coronary care unit, being mechanically ventilated with a positive end expiratory pressure greater than 5 cm H2O, with noncardiogenic pulmonary edema on chest x-ray within 48 hours of being noted to have a P/F ratio < 150.

Exclusion criteria includes patients < 18 years of age, patients for whom no aggressive measures are desired, patients who are already receiving "rescue methods" (prone positioning, advanced ventilator modes, paralytics), trauma patients, vulnerable patient groups (pregnant, prisoners), patients who have undergone a surgical operation during their time on the ventilator, patients with end stage liver disease, patients on chronic ventilators, and asthmatics.

Local Number of Subjects This study will seek to enroll 26 patients each in the treatment and control arm.

Study-Wide Number of Subjects This is a single center study. Study Timelines Plans will be to complete the study within 12 months from the time of start. Study Endpoints The patient is liberated from the ventilator, discharged from the ICU, discharged from the hospital, or dies.

Procedures Involved The only procedure involved would be the administration of N-acetylcysteine via nebulization, which would be administered to the patient by respiratory therapy in the dosage of 3 2 mL 20% solution acetylcysteine (or 6 4 mL of 10% solution) along with inhaled albuterol via endotracheal tube every six hours for 72 hours total. The control arm will have saline administered with the albuterol every six hours. Both arms will have additional bronchodilators administered as indicated clinically (bronchospasm, COPD, peak airway pressure elevation, etc.).

The patients would be monitored daily in the ICU setting with lab work, including arterial blood gases, chemistry panels, complete blood counts. They would have all routine critical care monitoring, such as hourly vital signs, urine output, ventilation parameters in accordance with the nature of their critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria includes adult patients admitted to the medical intensive care unit or coronary care unit, being mechanically ventilated with a positive end expiratory pressure greater than 5 cm H2O, with noncardiogenic pulmonary edema on chest x-ray within 48 hours of being noted to have a P/F ratio < 150.

Exclusion Criteria:

* Exclusion criteria includes patients < 18 years of age, patients for whom no aggressive measures are desired, patients who are already receiving "rescue methods" (prone positioning, advanced ventilator modes, paralytics), trauma patients, vulnerable patient groups (pregnant, prisoners), patients who have undergone a surgical operation during their time on the ventilator, patients with end stage liver disease, patients on chronic ventilators, and asthmatics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Ventilator days | From time of intubation until one of predefined endpoints (up to 60 days)
  Number of days requiring mechanical ventilation

SECONDARY OUTCOMES:
Mortality | up to 60 days
  Number of days until expiring
ICU days | From time of admission to the ICU until transfer out of the unit (up to 60 days)
  Number of days in the ICU
P/F ratio | Daily until the predefined endpoints (up to 60 days)
  A measure of the partial pressure of oxygen divided by the percentage of inhaled oxygen
Use of "rescue" maneuvers | Daily until the predefined endpoints (up to 60 days)
  Using airway pressure release ventilation, paralytics, or proning

CONTACTS AND LOCATIONS:
Overall Officials: Judson Lewis, MD, Principal Investigator — Prisma Health-Midlands
Locations (1):
- Palmetto Health Richland, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No